CLINICAL TRIAL: NCT04508894
Title: Ketamine Versus Dexmedetomidine as an Adjuvant in Ultrasound-guided Supraclavicular Brachial Plexus Block
Brief Title: Ketamine Versus Dexmedetomidine in Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 146:4/2019
Record Dates: First submitted 2020-08-02; First posted 2020-08-11 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Supraclavicular Brachial Plexus Block
MeSH Terms: interventions — Bupivacaine; Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Supraclavicular Brachial Plexus Block using 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline
  Interventions: Drug: Supraclavicular Brachial Plexus Block with bupivacaine
- Ketamine group (Active Comparator): Supraclavicular Brachial Plexus Block using 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline plus 1 mg\kg ketamine
  Interventions: Drug: Supraclavicular Brachial Plexus Block with Ketamine
- Dexmedetomidine group (Active Comparator): Supraclavicular Brachial Plexus Block using 20 ml 0.5% bupivacaine and 20 ml 0.9% normal saline plus 1µg\kg dexmedetomidine
  Interventions: Drug: Supraclavicular Brachial Plexus Block with Dexmedetomidine

INTERVENTIONS:
Drug: Supraclavicular Brachial Plexus Block with bupivacaine — drug: 20 ml 0.5%bupivacaine plus 20 ml 0.9% normal saline is administered around the brachial plexus on the operative side Drug: IM diclofenac sodium (75 mg amp) is injected if VAS more than 4.
  Device: ultrasound-guided supraclavicular Brachial Plexus nerve block
  Other Names: C group
  Arms: Control group
Drug: Supraclavicular Brachial Plexus Block with Ketamine — drug: 20 ml 0.5%bupivacaine, 20 ml 0.9% normal saline plus 1mg\kg ketamine is administered around the brachial plexus on the operative side Drug: IM diclofenac sodium (75 mg amp) is injected if VAS more than 4.
  Device: ultrasound-guided supraclavicular Brachial Plexus nerve block
  Other Names: K group
  Arms: Ketamine group
Drug: Supraclavicular Brachial Plexus Block with Dexmedetomidine — drug: 20 ml 0.5%bupivacaine, 20 ml 0.9% normal saline plus 1µg\kg dexmedetomidine is administered around the brachial plexus on the operative side Drug: IM diclofenac sodium (75 mg amp) is injected if VAS more than 4.
  Device: ultrasound-guided supraclavicular Brachial Plexus nerve block
  Other Names: D group
  Arms: Dexmedetomidine group

SUMMARY:
Intervention model description: The patients were randomly classified into three groups using computer-generated table numbers each contain (25) patients.

Ketamine group (group K): 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline plus 1 mg\kg ketamine, Dexmedetomidine group (group D): 20 ml 0.5% bupivacaine and 20 ml 0.9% normal saline plus 1µg\kg dexmedetomidine Control group (group C): 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline. Masking: double-blind (participant and investigator) Masking Description: The investigator's study is a prospective, randomized, double-blind

DETAILED DESCRIPTION:
This randomized, prospective, double-blind study was carried out on 75 ASA Physical Status I-II adults aged 18-75 years old scheduled to undergo elective and emergency forearm and hand surgeries under ultrasound-guided supraclavicular brachial plexus block. After obtaining the local ethics committee of El-Minia university hospital approval and written informed consent was taken of the patient, this study was conducted from April 2019 to February 2020 in El-Minia university hospital. The investigators excluded any patient with bleeding disorders, damage or disease of the brachial plexus, uncontrolled diabetes mellitus, and patients with neuromuscular diseases, Patients with a local skin infection at the site of injection or patients with known hypersensitivity to studied drugs.

Preoperative assessment and preparation: A careful assessment of medical history, general examination including chest, heart, abdomen, site of injection and other systems were carried out. Routine investigations were done as complete blood picture, ECG (electrocardiogram) renal and liver functions. An explanation of the visual analog scale was done to each patient.

Preparation of the studied medications: The patients were randomly classified into three groups using computer-generated table numbers each contains (25) patients. Ketamine group (group K): 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline plus 1 mg\kg ketamine, Dexmedetomidine group (group D) 20 ml 0.5% bupivacaine and 20 ml 0.9% normal saline plus 1µg\kg dexmedetomidine (precedex® Hospira,Inc., Lake Forest USA).

Control group (group C) 20 ml 0.5%bupivacaine and 20 ml 0.9% normal saline. All medications were prepared in similar sterile coated bottles by the supervisor who didn't include in the anesthetic or operative team, 75 bottles numbered from 1 to 75 were prepared. After completion of the study, the key was opened by the supervisor Block technique: On patient's arrival to the operating room, a 20 G intravenous cannula was inserted in a peripheral vein of unaffected limb and standard monitoring commenced as noninvasive blood pressure (NIBP), (ECG), and Oxygen saturation (Spo2) (UltraviewSL2700, Spacelaps, USA), all equipment and drugs for general anesthesia and resuscitation were prepared, the ultrasound device (Sonosite, Nanomax, USA ) lubricating gel, 21guge 50 mm length, short bevel, insulated stimulating needle (Laboratoires pharmaceutiques, Vygon, France). Patient lie supine with the head turned to the other side and ipsilateral arm adducted gently with a flexed elbow. Under the complete aseptic condition, the identified area and the ultrasound probe was prepared with anti-septic (Povidone-Iodine 10%) solution and the skin infiltrated with 1-2 ml of lidocaine 2% solution subcutaneously, the brachial plexus was visualized by placing the transducer in the sagittal plane in the supraclavicular fossa behind the middle-third of the clavicle. Two distinct appearances of the supraclavicular brachial plexus was seen, it either appeared as a grape-like cluster of 5 to 6 hypoechoic circles, located lateral and superior to the subclavian artery between the anterior and middle scalene muscles at the lower cervical region or as 3 hypoechoic circles with hyperechoic outer rings, the predetermined volume of 40 mL of the study drug solution was administered around the brachial plexus after negative aspiration to avoid accidental intravascular injection, expansion of the brachial plexus sheath was considered as an indication of correct needle placement, multiple injections were used to deposit the total amount of the study drugs, skin massage for about 3 minutes was done to facilitate drug distribution.

Parameters assessed:

* Hemodynamic data: The hemodynamic variables as HR, MAP and Spo2 were assessed. The parameters were recorded preoperatively just before the block as a baseline value, at 5,10,20,30,60, 90 minutes during the operative time and at 1,2,4,6,9 and 12 hours after the end of the operation.
* Sensory block was assessed by pinprick test using a 3-point scale [16] Grade 0 = normal sensation, Grade 1 = loss of sensation of pinprick (analgesia), and Grade 2 = loss of sensation of touch (anesthesia).
* Motor block was determined by thumb abduction (radial nerve), thumb adduction (ulnar nerve), thumb opposition (median nerve), and flexion of elbow (musculocutaneous nerve) according to the modified Bromage 3 point scale: Grade 0: Normal motor function with full flexion and extension of elbow, wrist, and fingers. Grade 1: Decreased motor strength with the ability to move the fingers only. Grade 2: Complete motor block with an inability to move the fingers [16].
* Onset time for sensory and motor block: the time interval between the end of local anesthetic administration and complete sensory and motor block by min.
* Sensory block duration: the time interval between the complete sensory block and complete resolution of anesthesia on all the nerves (score 0(
* Motor block duration: the time interval from complete motor block to complete recovery of motor function of hand and forearm (grade 0) by hours.
* Visual analog scale (VAS): postoperative, the patients were familiarized with a 10-point visual analog scale (VAS) ranged from 0 = no pain, up to 10 = the worse imaginable pain. VAS was measured at 1, 2, 3, 6, 9, 12 hours. When it equals or >4 the investigators give IM diclofenac sodium (75 mg amp) (Voltaren, Novartis Pharmaceuticals Corporation, Switzerland).
* Time of first analgesic request: The time passed from supraclavicular brachial plexus block to the patient's first request for analgesic medication by hours
* Total analgesic requirements in 24 hours) diclofenac consumption)
* Sedation score: was assessed according to the modified Ramsay Sedation Scale 1987(RSS) from 1-6 as follows: 1 = anxious, agitated, restless; 2 = cooperative, oriented, tranquil; 3 = responds to commands only; 4 = brisk response to light glabellar tap or loud noise; 5 = sluggish response to light glabellar tap or loud noise; 6 = no response [17].
* Adverse effects: any adverse effects such as hypotension (i.e. 20% decrease relative to baseline), bradycardia (HR <60 beats/min), nausea, vomiting, hypoxemia (SpO2 <90%), local hematoma, hemothorax, pneumothorax, recurrent laryngeal nerve block, intravascular injection, Horner's syndrome and signs of local anesthetic toxicity were recorded during the operation and for 12 hours postoperative.

ELIGIBILITY:
Inclusion Criteria:

* American Physical Status I or II
* patients undergoing elective and emergency forearm and hand surgeries

Exclusion Criteria:

* Patient with bleeding disorders
* Damage or disease of the brachial plexus
* Uncontrolled diabetes mellitus
* Patients with neuromuscular diseases
* Patients with a local skin infection at the site of injection
* Patients with known hypersensitivity to studied drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate duration of sensory block | 24 hours after block
  Sensory block duration: the time interval between the complete sensory block and complete resolution by hours

SECONDARY OUTCOMES:
Evaluate onset of sensory and motor block | 30 minute after block
  Onset time for sensory and motor block: the time interval between the end of local anesthetic administration and complete sensory and motor block by min.
Assess postoperative pain score | For 24 hours after surgery
  The severity of postoperative pain will be measured and recorded by using the visual analogue scale (VAP) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
time to first analgesic request | 24 hours
  Time for the first request to rescue analgesia (in hours)
total analgesic requirements | 24 hours after surgery
  Total diclofenac consumption requirements in 24 hours
sedation score | 24 hours after surgery
  Ramsay Sedation Scale from 1-6 as follows: 1 = anxious, agitated, restless; 2 = cooperative, oriented, tranquil; 3 = responds to commands only; 4 = brisk response to light glabellar tap or loud noise; 5 =sluggish response; 6 = no response

CONTACTS AND LOCATIONS:
Overall Officials: Haidy S Mansour, MD, Principal Investigator — assistant professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Minya University, Minya, Egypt

DOCUMENTS (1):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT04508894/Prot_000.pdf